CLINICAL TRIAL: NCT05892146
Title: Strategy Therapy on Early Phase Cancer Therapeutics-Related Cardiac Dysfunction Patients
Brief Title: Strategy Therapy on Cancer Therapy-Related Cardiac Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Ping-Yen Liu, Doctor/Professor, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: A-BR-110-021
Record Dates: First submitted 2023-05-26; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Chemotherapeutic Toxicity; Cardiotoxicity; Heart Failure; Breast Cancer; Lymphoma
MeSH Terms: conditions — Cardiotoxicity; Heart Failure; Breast Neoplasms; Lymphoma | interventions — Secondary Prevention

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Prevention therapy (Experimental): Sacubitril/Valsartan (25/80) mg twice a day for 1 year
  Interventions: Drug: Prevention therapy
- Conventional therapy (No Intervention): No intervention
- Global longitudinal strain (GLS) function decreased >15%, No intervention (No Intervention): With the value of GLS function via echocardiography study decreased >15%, No intervention
- GLS function descending >15%, Rescue therapy (Experimental): Sacubitril/Valsartan (25/80) mg twice a day for 1 year
  Interventions: Drug: Rescue therapy

INTERVENTIONS:
Drug: Prevention therapy — Sacubitril/Valsartan (25/80) mg twice a day for 1 year
  Arms: Prevention therapy
Drug: Rescue therapy — Sacubitril/Valsartan (25/80) mg twice a day for 1 year
  Arms: GLS function descending >15%, Rescue therapy

SUMMARY:
The investigators use the cancer registration system of National Cheng Kung University Hospital to timely screen and evaluate those patients having breast cancer or lymphoma to enroll patients to participate in this clinical trial. The investigators planned an earlier initiation of Sacubitril/Valsartan treatment on breast cancer and lymphoma patients before the chemotherapy, and starting therapeutic intervention by Sacubitril/Valsartan once the heart damage sign appeared via novel echocardiography. The investigators aim to assess the protective and therapeutic benefit of cardioprotective drugs on the cardiotoxicity of anti-cancer therapy.

DETAILED DESCRIPTION:
The investigators use the cancer registration system of National Cheng Kung University Hospital to timely screen and evaluate those patients having breast cancer or lymphoma to enroll patients to participate in this clinical trial. Also, the Patient Recruitment System support to complete the patients' database. The investigators cooperate with other hospitals in South Taiwan to carry on an early phase clinical trial, named "Strategy by novel anti-heart failure therapy on early phase Cancer Therapeutics-Related Cardiac Dysfunction (CTRCD) patients" focusing on the either preventive strategy to earlier initiation of Sacubitril/Valsartan treatment on breast cancer and lymphoma patients before the chemotherapy, and starting therapeutic intervention by Sacubitril/Valsartan once the heart damage sign appeared via novel echocardiography, and collect clinical and genetic information from the enrolled patients. These patients randomized into 2 groups: cardioprotective drug vs. placebo. The regular assessment of cardiac function is as following: baseline (prior to anti-cancer treatment) and every 3 months. Thereafter. The investigators aim to assess the protective and/or therapeutic benefit of cardioprotective drugs on the cardiotoxicity of anti-cancer therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are newly diagnosed with breast cancer or lymphoma and never accepted anti-cancer therapy
* Age 20-65 years old
* Systolic blood pressure ≥ 110 mmHg

Exclusion Criteria:

* End-stage renal disease (estimated Glomerulus Filtration Rate <15 mL/min/1.73 m2)
* Echocardiography Baseline left ventricle ejection fraction < 50%
* Allergy history to angiotensin receptor blockers
* Life expectancy < 1 year
* Pregnancy
* Unwilling to participate in this clinical study

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in absolute global longitudinal strain value measured by left ventricular global peak systolic longitudinal strain | 1 year
  Left ventricular global peak systolic longitudinal strain by cardiac echo

SECONDARY OUTCOMES:
Change in left ventricular ejection fraction value measured by echocardiography | 1 year
  Left ventricular ejection fraction by cardiac echo
Heart failure hospitalization | 1 year
  admission due to heart function deterioration
All-cause mortality | 1 year
  All types of death
Change in cardiac biomarkers: including N terminal pro B type natriuretic peptide (NT-proBNP) and high-sensitivity cardiac Troponin (hs-cTnT) | 1 year
  Cardiac biomarkers (NT-proBNP and hs-cTnT) changes

CONTACTS AND LOCATIONS:
Overall Officials: Ping-Yen Liu, MD, PhD, Principal Investigator — National Cheng Kung University Hospital, Tainan, Taiwan
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No